CLINICAL TRIAL: NCT06444867
Title: An Open-label, Phase 1b, Multi-site Trial to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Following a Single Dose of LEO 158968 in Subjects With Gout Flares
Brief Title: A Study to Evaluate Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of LEO 158968
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0189-2318; 2023-508793-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Joint Pain; Gout Flares; Joint Inflammation
Keywords: LEO 158968
MeSH Terms: conditions — Arthralgia; Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEO 158968 (Experimental): Participants with gout flares will receive a single SC dose of LEO 158968 on Day 1.
  Interventions: Drug: LEO 158968

INTERVENTIONS:
Drug: LEO 158968 — SC injection

SUMMARY:
The main objective of the study is to evaluate the effect on pain of a single, subcutaneous (SC) dose of LEO 158968 in participants with gout flares.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained prior to any protocol-related procedures.
* Participants meeting the American College of Rheumatology (ACR/EULAR) 2015 gout criteria with a score ≥8.
* Presence of a gout flare for no longer than 96 hours prior to the baseline visit.
* In case of naïve or newly diagnosed participants, the presence of monosodium urate (MSU) crystals in synovial fluid will be evaluated and confirmed.
* At least 1 joint affected by acute gout (eg, ankle, foot, knee, toe). Participants may have oligoarticular gout, defined as >1 and <5 affected joints. However, participants with polyarticular gout are not eligible. In case the participant has more than one affected joint, the investigator should select the most symptomatic joint (most painful/with more inflammatory signs) for the study assessments (primary endpoint), and it will be identified as the 'index joint'.
* At screening and baseline (Day 1), a participant-reported joint pain at rest of ≥50 mm on a 0-100 mm VAS with pain intensity ≥2 using a 5-point Likert scale and at least 2 of the following criteria in the target joint:

  1. participant-reported flare.
  2. participant-reported warm joint.
  3. participant-reported swollen joint.
* Body mass index: ≤40 kg/m², at screening.
* Participants on ULT (xanthine oxidase inhibitors, uricosuric agents) with no changes in therapy for at least 2 weeks before dosing.
* Male participants, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from admission to the clinical research center until all follow-up procedures are complete. Adequate contraception for the male participant (and his female partner, if she is of childbearing potential) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence from heterosexual intercourse, in accordance with the lifestyle of the participant, is also acceptable.
* Participants with hypertension, cardiovascular disease, diabetes, or renal disorder are required to be on a stable dose and schedule, with no changes in therapy for at least 4 weeks before screening and baseline, are expected to remain on a stable regimen during trial participation, and the diseases are biologically and clinically controlled.

Exclusion Criteria:

* Use of specified pain relief medications, including systemic glucocorticoids, within 4 weeks before the baseline visit, and weak and strong opioids, colchicine, and nonsteroidal anti inflammatory drugs within 7 days before the baseline visit.
* Presence of an acute gout flare in more than 4 joints at the baseline visit.
* Received a live vaccine within 4 weeks before dosing or receiving a live vaccine during the trial.
* Other causes of acute or chronic inflammatory arthritis (including rheumatoid arthritis, psoriatic arthritis, and calcium pyrophosphate deposition disease), tophaceous gout, or evidence/suspicion of infectious/septic arthritis.
* History of malignancy within the past 5 years, with the exception of basal cell skin cancer, carcinoma-in-situ of the cervix, or low-risk prostate cancer after curative therapy.
* Known hypersensitivity to any components of the product.
* Presence of active or recurrent bacterial, fungal, or viral infections within 15 days prior to the baseline visit, or presence of human immunodeficiency virus (HIV) infection, and hepatitis B and C infection.
* Presence of active or latent tuberculosis (to be determined by chest X-ray and a tuberculosis screening questionnaire).
* Uncontrolled clinically significant hematologic, pulmonary, endocrine, metabolic, gastrointestinal, central nervous system, or hepatic disease.
* Unstable cardiovascular disease, defined as a recent clinical deterioration (eg, unstable angina, myocardial infarction, cerebrovascular events, or rapid atrial fibrillation) in the last 3 months prior to screening, or a cardiac hospitalization within the 3 months prior to screening.
* Participants who have undergone major surgery within 2 weeks before the baseline visit or have an unhealed operation wound.
* The presence of any medical or psychological condition or laboratory results that, in the Investigator's opinion, might create a risk to the participants or the trial.
* History of alcohol or substance abuse within the 12 months prior to the baseline visit or any condition associated with poor compliance as judged by the Investigator.
* Clinically significant general pain or non-gout-related joint pain that would interfere with the participant's ability to accurately assess pain in the target joint, at the discretion of the Investigator.
* Current participation in any other interventional clinical trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Patient-reported Pain Intensity Score of 0 or 1 as Assessed by the 5-point Likert Scale on Day 4 | Day 4
  The 5-point Likert scale for pain intensity assesses the degree of pain experienced by a participant. The scale is scored from 0 (no pain) to 4 (severe pain).

SECONDARY OUTCOMES:
Number of Participants with a Patient-reported Pain Intensity Score of 0 or 1 as Assessed by the 5-point Likert Scale on Day 8 | Day 8
  The 5-point Likert scale for pain intensity assesses the degree of pain experienced by a participant. The scale is scored from 0 (no pain) to 4 (severe pain).
Number of Participants with a ≥2-point Reduction in Patient-reported Pain Intensity Score as Assessed by the 5-point Likert | Day 1 to Day 8
  The 5-point Likert scale for pain intensity assesses the degree of pain experienced by a participant. The scale is scored from 0 (no pain) to 4 (severe pain).
Number of Participants Experiencing a Change in Pain Intensity in Affected Joints as Assessed by the Visual Analog Scale (VAS) Pain Score | Baseline to Day 8
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Baseline to Day 85
  A TEAE is defined as any event not present prior to administration of the trial drug or any event already present that worsens in either severity or frequency following exposure to the trial drug. A serious AE (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires participant to be hospitalized, results in disability, is a congenital anomaly, is a medical condition not immediately life-threatening but that requires intensive treatment in emergency room or at home. Any clinically significant changes in physical examination findings and abnormal objective test findings (eg, laboratory, x-ray, ECG) will be recorded as AEs.
Number of Participants with LEO 158968 Anti Drug Antibodies (ADA) from Baseline to Day 85 | Baseline to Day 85
Number of Participants with LEO 158968 ADA from Baseline to Day 29 | Baseline to Day 29
Number of Participants Using Rescue Medications from Baseline to Day 8 | Baseline to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (3):
- LEO Pharma Investigational Site, Lille, France
- LEO Pharma Investigational Site, Venlo, Netherlands
- LEO Pharma Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No